CLINICAL TRIAL: NCT00189475
Title: A Pilot Study to Evaluate the Potential of Montelukast to Prevent the Development of Nasal Symptomatology During Natural Viral Upper Respiratory Infections
Brief Title: Evaluate the Potential of Montelukast to Prevent Nasal Symptomatology During Colds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deborah Gentile (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Deborah Gentile, Physician , Allergy and Asthma Institute, West Penn Allegheny Health System
Organization: West Penn Allegheny Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC - 3559
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Upper Respiratory Infection
Keywords: Cold; Upper Respiratory Infection
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Active Comparator): Treated for 4 months with montelukast 4 mg per day
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): Treated for 4 months with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast
  Arms: Montelukast
Drug: Placebo
  Arms: Placebo

SUMMARY:
Assesses the efficacy of treatment with montelukast 10 mg PO QD x 5 days versus placebo for the treatment of viral-induced upper respiratory infection in healthy adults aged 18-50 years.

DETAILED DESCRIPTION:
This is a randomized double-blinded placebo controlled trial to assess the efficacy of treatment with montelukast 10 mg PO QD x 5 days versus placebo for the treatment of viral-induced upper respiratory infection in healthy adults aged 18-50 years. All subjects complete daily assessments of cold symptoms, nasal clearance rates and secretion rates during each day of the study. Phlebotomy is performed once for the determination of cytokine genotyping and allergy skin testing is performed once for the assessment of atopy.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 50 years of age.
* Male or female, who are not pregnant or lactating.
* Common cold symptoms for less than 24 hours.
* At least 2 of the following 9 symptoms: cough, headache, hoarseness, muscle ache, nasal drainage, nasal congestion, scratch throat, sneezing and malaise.

Exclusion Criteria:

* Investigational medication in past 30 days.
* Known hypersensitivity to any ingredients in study medication.
* History of asthma or other chronic diseases.
* Females of childbearing potential who are not using a medically acceptable form of birth control.
* Patients with nasal ulcers within the past 1 month, nasal surgery within the past 6 months, nasal trauma within the past 2 months or presence of nasal polyps or nasal deformities causing significant nasal obstruction.
* Females with a positive urinary HCG test.
* Patients with a positive rapid antigen test for streptococcal infection.
* Common cold symptoms for more than 24 hours.
* Patients who are users of illicit drugs.
* Patients who are on rifampin or phenobarbital.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2003-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Gentile, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Montelukast: Treated for 4 months with montelukast 4 mg per day
  Montelukast
Period: Overall Study
Arm/Group | Montelukast | Placebo
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast | Placebo | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 42 | 84
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Male | 13 | 13 | 26
  Female | 29 | 29 | 58
Region of Enrollment [Number; unit: participants] — All subjects were enrolled through the Asthma and Allergy Dept at West Penn Allegheny Health System.
  participants
    United States | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Nasal Secretion Weights
Time Frame: 6 days after naturally acquiring an upper respiratory infection
Measure: Mean (Standard Error); unit: grams
Groups:
- Montelukast: Montelukast 10mg per day for 6 days
- Placebo: Treated for 6 days with placebo
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 42 | 42
grams
  Day 1 | 3.5 (0.4) | 4.2 (0.6)
  Day 6 | 1.2 (0.4) | 2.6 (0.4)

ADVERSE EVENTS:
Arm/Group | Montelukast | Placebo
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No